CLINICAL TRIAL: NCT05972850
Title: Vivo Heart: Home-Based Virtual Exercise Program for Older Adults With Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00094007; P30AG021332 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Disease
Keywords: home-based cardiac rehabilitation; mobile health technologies; strength and physical function; synchronous virtual exercise program
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 40 rural-living older adults (60-80 years) with a history of cardiovascular disease (prior myocardial infarction, angina, or coronary procedure) who are medically cleared for exercise by their cardiologist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vivo Heart (Experimental): This virtual intervention will include weekly group exercise sessions with a Vivo trainer (2 times/week), weekly health education classes with a registered dietitian (RD) (1 time/week), and two individual meetings with the RD over the course of 12 weeks. Participants will also be asked to complete a weekly aerobic exercise session on their own (1 time/week).
  Interventions: Behavioral: Vivo Heart

INTERVENTIONS:
Behavioral: Vivo Heart — Vivo is an online, live, small group fitness program developed for older adults that uses individually tailored dual-tasked (i.e., cognitive-motor) exercises to improve strength, endurance, balance, and cognition and incorporates social engagement. Certified trainers deliver instruction and coaching through an interactive session for 45 min, 2-3 times/week.
  Other Names: Vivo

SUMMARY:
This pilot study will assess the feasibility and generate preliminary efficacy data of a novel, synchronous, home-based exercise training program for rural older adults with cardiovascular disease (CVD) using Vivo, an online, live, small group fitness program developed for older adults. It uses individually tailored dual-tasked (i.e., cognitive-motor) exercises to improve strength, endurance, balance, and cognition and incorporates social engagement. Certified trainers deliver instruction and coaching through an interactive session (45 min, 2-3 times/week) delivered over 12 weeks. Vivo Heart adapts this unique program to meet the cardiac rehabilitation needs of older adults with CVD. The specific aims are to evaluate the feasibility, acceptability, and uptake of Vivo Heart (Aim 1) and obtain pre- and post-intervention measures of exercise capacity, strength, lower-extremity physical function, cognition, quality of life, stress, fatigability, physical activity, and aging biomarkers (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* 60 - 80 years
* Lives in a rural area based on established urban-rural definitions (e.g., RUCA codes, RUCC, UIC)
* A qualifying Cardio Vascular Disease (CVD) event or procedure
* Cognitively unimpaired Telephone Interview for Cognitive Status (TICS-m ≥32)
* No major depressive symptoms Patient Health Questionnaire (PHQ-8 <10)
* Ambulatory and community-dwelling
* Less than 150 min per week of moderate-to-intensive aerobic or resistance exercise in the past month
* Medically cleared for exercise if event was within the last 6 months
* Access to a tablet or computer and internet/Wi-Fi in defined exercise space
* Able to provide own transportation to study visits
* Not participating in a clinical trial
* Willing to provide informed consent

Exclusion Criteria:

* <60 years or >80 years
* Lives in non-rural area
* No CVD or a qualifying event or procedure
* Dementia or severe cognitive impairment (TICS-m <32)
* Clinical depression (PHQ-8 ≥10)
* Non-ambulatory, institutionalized, or requires walker
* Regular aerobic or resistance exercise (including current participation in a cardiac rehab program)
* Not medically cleared for exercise
* Advanced kidney disease requiring dialysis or dialysis anticipated within 6 months
* Insulin-dependent diabetes
* Use of any supplemental oxygen for COPD
* Significant impairment from a prior stroke
* Progressive neurologic disease (Parkinson's, ALS, multiple sclerosis, Alzheimer's disease, dementia)
* Severe arthritis, fracture, chronic injury, or other musculoskeletal disorder that prevents walking independently
* Cancer (not including non-melanoma skin cancers) requiring treatment with the past year
* Excessive alcohol consumption (>7/week alcoholic beverages for women and >14/week for men) in the past month
* Joint replacement or other orthopedic surgery in past 12 months or planned in next 6 months
* No computer, tablet or internet access
* No access to transportation for travel to study visits
* Current participation in a clinical trial
* Inability or unwillingness to comply with the study requirements

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Completion Rate | Week 12
  Completion rate which will be determined by the percentage of enrolled participants who complete the study with ≥80% compliance.

SECONDARY OUTCOMES:
Recruitment Rate | Year 1
  Recruitment rate will be determined by the total number of enrolled participants divided by the number of months recruitment occurred.
Recruitment Yield | Year 1
  Recruitment yield will be determined based on the number of participants randomized relative to the total number of volunteers screened
Compliance Rate | Week 12
  Compliance will be determined based on adherence to the prescribed intervention. Compliance metrics will include attendance at the exercise sessions, health education classes, and dietary counseling sessions.
Retention Rate | Week 12
  Retention will be determined by the percentage of enrolled participations who complete follow-up testing.
Satisfaction Survey Scores | Week 12
  Acceptability will be assessed at the end of the study using a program satisfaction survey.
Continuation Rate | Year 1
  Uptake will be determined by the number of participants who continue in the Vivo program after the study is over.

OTHER OUTCOMES:
VO2 peak | Week 12
  Change in VO2 peak
Montreal Cognitive Assessment (MoCA) | Week 12
  Change in overall cognition (0-30)
Digit Symbol Coding (DSC) | Week 12
  Change in processing speed, working memory, visuospatial processing, and attention (secs)
Timed Up and Go (TUG) | Week 12
  Change in time to complete (secs)
Expanded Short Physical Performance Battery (eSPPB) | Week 12
  Change in score (0-4)
The Four Square Step Test (FSST) | Week 12
  Change in time to complete (secs)
4-step Stair Climb Test (4SCT) | Week 12
  Change in time to complete (secs)
Grip Strength | Week 12
  Change in grip strength (kg)
Perceived Stress Scale (PSS) | Week 12
  Change in score
Short Form-36 Health Survey (SF-36) | Week 12
  Change in score
UCLA Loneliness Scale | Week 12
  Change in score
Life Space | Week 12
  Change in score
Pittsburgh Fatigability Scale (PFS) | Week 12
  Change in score
Blood pressure | Week 12
  Change in systolic and diastolic blood pressure (mmHg)
Heart rate | Week 12
  Change in resting heart rate (bpm)

CONTACTS AND LOCATIONS:
Overall Officials: Tina E Brinkley, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT05972850/ICF_000.pdf